CLINICAL TRIAL: NCT07274488
Title: The Effect of Preoxygenation on Gastric Decompression in Laparoscopic Cholecystectomies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: EBRU-YURDAKUL-VURAL-ANKARA-001
Record Dates: First submitted 2025-11-19; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Cholelithiasis
Keywords: Laparoscopic Cholecystectomy; Preoxygenation; Gastric Decompression; Gastric Insufflation; Postoperative Sore Throat; Orogastric tube
MeSH Terms: conditions — Cholelithiasis

STUDY DESIGN:
Intervention Model Description: Prospective, Randomized, Single-Blind Clinical Trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ventilation Group (Group A) (Active Comparator): Patients who underwent mask ventilation after anaesthesia induction (Group A, n=64)
  Interventions: Procedure: Mask Ventilation
- Preoxygenation Group (Group B) (Experimental): Those preoxygenated until their end-tidal oxygen (EtO₂) level exceeded 85% and not ventilated with a mask before induction (Group B, n=64)
  Interventions: Procedure: Preoxygenation

INTERVENTIONS:
Procedure: Preoxygenation — Patients in the preoxygenation group were preoxygenated prior to induction until EtO₂ >85%, and patients were intubated without mask ventilation.
  Arms: Preoxygenation Group (Group B)
Procedure: Mask Ventilation — After anaesthesia induction, mask ventilation is administered until intubation, and preoxygenation is not performed.
  Arms: Ventilation Group (Group A)

SUMMARY:
Aim: Gastric insufflation caused by mask ventilation during laparoscopic surgeries may affect the surgical field, lead to regurgitation of gastric contents, and consequently cause aspiration pneumonia. In this study, we aimed to investigate the effect of preoxygenation instead of mask ventilation in laparoscopic cholecystectomies (LC) on the need for decompression due to gastric insufflation, as well as its impact on postoperative sore throat and the presence of bleeding in aspiration in patients requiring an orogastric (OG) tube.

Materials and Methods: This single-center, prospective, observational study included 128 patients aged 18-65 years with ASA I-III undergoing LC surgery. After anesthesia induction, patients were divided into two groups: those ventilated with a mask (Group A, n=64) and those preoxygenated until their end-tidal oxygen (EtO₂) level exceeded 85% and not ventilated with a mask before induction (Group B, n=64). Anesthesia induction was performed in a standardized manner with appropriate doses for each patient. After administration of a muscle relaxant, patients were intubated by the same anesthesiologist following a 2-minute waiting period. The development of gastric insufflation, the need for OG tube placement, sore throat, and the presence of bleeding in aspiration were compared between the groups.

DETAILED DESCRIPTION:
Exclusion criteria for participation in the study:

* Age under 18 or over 65 years,
* Patients who do not wish to participate in the study,
* Patients classified as ASA IV or V,
* History of difficult intubation.

Criteria for termination of study participation:

* Failure to perform endotracheal intubation on the first attempt
* Presence of difficult intubation
* Occurrence of oropharyngeal or laryngeal trauma during intubation

Expected Benefits and Risks of the Study:

We hypothesize that in the operating rooms of the Oncology Hospital at Ankara City Hospital, Ministry of Health of the Republic of Türkiye, preoxygenation instead of mask ventilation during general anesthesia for laparoscopic cholecystectomies may reduce gastric insufflation, potentially improve surgical comfort, and have a positive effect on postoperative sore throat caused by swallowing, since the use of orogastric tubes may no longer be necessary.

ELIGIBILITY:
Inclusion Criteria:

Scheduled to undergo laparoscopic cholecystectomy under general anesthesia

* Patients aged 18-65 years
* ASA physical status I, II, or III

Exclusion Criteria:

* Patients younger than 18 years or older than 65 years
* ASA physical status IV or V
* History of difficult intubation

Termination Criteria:

* Failure to achieve successful intubation on the first attempt
* Difficult intubation during the procedure
* Oropharyngeal or laryngeal trauma occurring during endotracheal intubation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Presence of Gastric Insufflation | Immediately after creation of pneumoperitoneum
  The surgeon assessed the degree of gastric distension after trocar placement and creation of pneumoperitoneum with CO₂. If gastric insufflation was present, an orogastric (OG) tube was inserted in both groups.

SECONDARY OUTCOMES:
Severity of Postoperative Sore Throat | Postoperative 10 minutes
  After extubation, patients who were transferred to the postoperative recovery unit were asked about the presence and severity of sore throat during swallowing. Sore throat was scored as follows:
  0 = no sore throat
  1. = mild sore throat
  2. = moderate sore throat
  3. = severe sore throat
Presence of Blood During Suction at Extubation | During extubation
  The presence of blood during oropharyngeal suction was recorded at the time of extubation in both groups. The relationship between the use of an orogastric (OG) tube and the presence of blood during suction was evaluated.
Postoperative presence of a blood smell in the mouth | Postoperative 10 minutes
  The presence of a blood smell in the mouth was assessed in the postoperative recovery unit after extubation. Patients were asked whether they noticed a blood smell in the oral cavity during the early postoperative period.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences (SBÜ) Ankara Bilkent City Hospital, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/36581835/
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC10510126/